CLINICAL TRIAL: NCT04464694
Title: Prospective, Single-blind, Randomised, Controlled, Multi-centre Study to Evaluate the Benefit of Ranibizumab as an Adjunctive Therapy to Vitrectomy for Patients With Proliferative Diabetic Retinopathy Combined With Diabetic Macular Oedema
Brief Title: Pre-vitrectomy Intravitreal Ranibizumab for Patients With Proliferative Diabetic Retinopathy Combined With Diabetic Macular Edema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-20-011
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Proliferative Diabetic Retinopathy; Diabetic Macular Edema
Keywords: PDR; DME; ranibizumab; vitrectomy
MeSH Terms: interventions — Ranibizumab; salicylhydroxamic acid; Vitrectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab (Experimental): Single intravitreal injection of ranibizumab (0.5 mg) 3~7 days before vitrectomy
  Interventions: Drug: Ranibizumab; Procedure: Pars plana vitrectomy
- Sham injection (Sham Comparator): Sham injection 3~7 days before vitrectomy
  Interventions: Other: Sham injection; Procedure: Pars plana vitrectomy

INTERVENTIONS:
Drug: Ranibizumab — Patients will receive single intravitreal injection of Ranibizumab 0.5 mg 3~7 days before vitrectomy.
  Other Names: Lucentis
  Arms: Ranibizumab
Other: Sham injection — Patients will receive single sham injection 3~7 days before vitrectomy.
  Arms: Sham injection
Procedure: Pars plana vitrectomy — Surgical procedure to remove the intravitreal hemorrhage and fibrosis membrane, and re-attach the retina, and perform endo laser photocoagulation on retina
  Other Names: Vitrectomy

SUMMARY:
To investigate ranibizumab's benefit on prevention of early postoperative vitreous haemorrhage in PDR-DME patients receiving vitrectomy.

DETAILED DESCRIPTION:
Primary Objective: To investigate ranibizumab's benefit on prevention of early postoperative vitreous haemorrhage in PDR-DME patients receiving vitrectomy.

Secondary Objective:To investigate ranibizumab's additional benefit on visual improvement, facilitation of surgery and postoperative outcomes in PDR-DME patients receiving vitrectomy.

Study design: This study is a prospective, randomized, single-blinded, blank-controlled, multi-center clinical trial that requires vitrectomy for PDR-DME patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old;
2. Type I or II diabetes mellitus, clinically diagnosed as diabetic macular edema
3. Diagnosed as proliferative diabetic retinopathy and pas plana vitrectomy (PPV) is required to undergo due to non-absorbent vitreous hemorrhage (VH), fibrovascular proliferation with vitreoretinal adhesions or tractional retinal detachment (TRD); or active severe proliferative retinopathy not responding to previous panretinal laser photocoagulation; as well as other indications of PPV at the investigator's discretion
4. Ability to provide written informed consent and comply with study assessments for the full duration of the study.

Exclusion Criteria:

1. Pregnancy or lactation;
2. History of stroke, peripheral vascular disease, angina or myocardial infarction within six months
3. Intraocular treatment with corticosteroids, anti-vascular endothelium growth factor or intraocular surgery within 45 days preceding baseline;
4. Clinically confirmed intraocular pressure (IOP) >=21 mmHg, uncontrolled glaucoma or iris neovascularization in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Early postoperative vitreous haemorrhage | From day 1 to week 4 after the vitrectomy
  To compare the incidence of the early postoperative vitreous haemorrhage between two arms

SECONDARY OUTCOMES:
Mean Best-corrected visual acuity (BCVA) at Month 3 | Month 3 after vitrectomy
  To compare the changes from baseline BCVA to mean BCVA at month 3 between two arms.
Mean Best-corrected visual acuity (BCVA) at Month 6 | Month 6 after vitrectomy
  To compare the changes from baseline BCVA to mean BCVA at month 6 between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Peiquan Zhao, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Ningbo Eye Hospital, Ningbo, Zhejiang
  - Eye & Ent Hospital of Fudan University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai JiaoTong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lo WR, Kim SJ, Aaberg TM Sr, Bergstrom C, Srivastava SK, Yan J, Martin DF, Hubbard GB 3rd. Visual outcomes and incidence of recurrent vitreous hemorrhage after vitrectomy in diabetic eyes pretreated with bevacizumab (avastin). Retina. 2009 Jul-Aug;29(7):926-31. doi: 10.1097/IAE.0b013e3181a8eb88. PMID 19584650
- [Result] Zhao LQ, Zhu H, Zhao PQ, Hu YQ. A systematic review and meta-analysis of clinical outcomes of vitrectomy with or without intravitreal bevacizumab pretreatment for severe diabetic retinopathy. Br J Ophthalmol. 2011 Sep;95(9):1216-22. doi: 10.1136/bjo.2010.189514. Epub 2011 Jan 27. PMID 21278146
- [Result] Comyn O, Wickham L, Charteris DG, Sullivan PM, Ezra E, Gregor Z, Aylward GW, da Cruz L, Fabinyi D, Peto T, Restori M, Xing W, Bunce C, Hykin PG, Bainbridge JW. Ranibizumab pretreatment in diabetic vitrectomy: a pilot randomised controlled trial (the RaDiVit study). Eye (Lond). 2017 Sep;31(9):1253-1258. doi: 10.1038/eye.2017.75. Epub 2017 May 12. PMID 28498374